CLINICAL TRIAL: NCT02142504
Title: Phase II, Randomized, Placebo-controlled, Double-blind, Safety and Immunogenicity Trial of Intramuscular Norovirus GI.1/GII.4 Bivalent Virus-Like Particle Vaccine in Healthy Adults
Brief Title: Safety and Immunogenicity of Norovirus Bivalent Virus-Like Particle Vaccine in Healthy Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NOR-201; U1111-1155-8803 (Other: World Health Organization)
Record Dates: First submitted 2014-05-09; First posted 2014-05-20 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Norovirus Prevention
Keywords: Drug therapy
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- GI.1/GII.4 15/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL) (Experimental): Intramuscular (IM) norovirus bivalent virus like particle (VLP) vaccine (15 µg of GI.1 norovirus VLP and 50 µg GII.4 norovirus VLP) adjuvanted with 50 µg monophosphoryl lipid A (MPL) and 500 µg aluminum hydroxide, on Day 1, followed by IM norovirus bivalent VLP vaccine (15 µg of GI.1 norovirus VLP and 15 µg GII.4 norovirus VLP) adjuvanted with 500 µg aluminum hydroxide (no MPL), on Day 365.
  Interventions: Biological: Norovirus Bivalent VLP Vaccine
- GI.1/GII.4 50/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL) (Experimental): IM norovirus bivalent VLP vaccine (50 µg of GI.1 norovirus VLP and 50 µg GII.4 norovirus VLP) adjuvanted with 50 µg monophosphoryl lipid A (MPL) and 500 µg aluminum hydroxide, on Day 1, followed by IM norovirus bivalent VLP vaccine (15 µg of GI.1 norovirus VLP and 15 µg GII.4 norovirus VLP) adjuvanted with 500 µg aluminum hydroxide (no MPL), on Day 365.
  Interventions: Biological: Norovirus Bivalent VLP Vaccine
- Saline Placebo + GI.1/GII.4 15/15 μg (No MPL) (Placebo Comparator): IM saline placebo on Day 1, followed by IM norovirus bivalent VLP vaccine (15 µg of GI.1 norovirus VLP and 15 µg GII.4 norovirus VLP ) adjuvanted with 500 µg aluminum hydroxide (no MPL), on Day 365.
  Interventions: Biological: Norovirus Bivalent VLP Vaccine; Drug: Placebo (Saline)

INTERVENTIONS:
Biological: Norovirus Bivalent VLP Vaccine — Norovirus GI.1/GII.4 bivalent VLP vaccine adjuvanted with or without MPL and/or aluminum hydroxide IM injection
Drug: Placebo (Saline) — Placebo-matching norovirus bivalent VLP vaccine
  Arms: Saline Placebo + GI.1/GII.4 15/15 μg (No MPL)

SUMMARY:
The purpose of this study is to evaluate the safety of the norovirus bivalent virus-like particle (VLP) vaccine for further development by assessing the rates of serious adverse events (SAEs), unsolicited adverse events (AEs), solicited local and solicited systemic AEs, Adverse Events of Special Interest (AESIs) and AEs leading to participant's withdrawal from the trial.

DETAILED DESCRIPTION:
The vaccine being tested in this study is called norovirus GI.1/GII.4 bivalent virus-like particle (VLP) vaccine adjuvanted with or without monophosphoryl lipid A (MPL) and with aluminum hydroxide. The norovirus vaccine is being tested to provide additional safety and immunogenicity data to enable the vaccine to be further developed. This study will look at the side effects in people who take different formulations of the norovirus vaccine.

The study will enroll approximately 450 participants. Participants will be randomly assigned (by chance, like flipping a coin) to one of the 3 treatment groups-which will remain undisclosed to the participant and study doctor during the study (unless there is an urgent medical need):

* one dose of GI.1/GII.4 (15 µg/50 µg) adjuvanted with MPL (50 µg) and aluminum hydroxide (500 µg) on Day 1 followed by one dose of GI.1/GII.4 (15 µg/15 µg) adjuvanted with aluminum hydroxide (500 µg) (without MPL) on Day 365
* one dose of GI.1/GII.4 (50 µg/50 µg) adjuvanted with MPL (50 µg) and aluminum hydroxide (500 µg) on Day 1 followed by one dose of GI.1/GII.4 (15 µg/15 µg) adjuvanted with aluminum hydroxide (500 µg) (without MPL) on Day 365
* one dose of Saline Placebo (dummy inactive injection) - this is a liquid that has no active ingredient-on Day 1 + GI.1/GII.4 (15 µg/15 µg) adjuvanted with aluminum hydroxide (500 µg) (without MPL) as primary vaccination on Day 365

All participants will be administered vaccine or placebo on Day 1 of the study and will receive a vaccination dose (reduced antigen content) of the norovirus vaccine on Day 365. Participants will be asked to record any symptoms that may be related to the vaccine or the injection site in a diary card for 7 days after each vaccination.

This multi-center trial will be conducted in the United States. The overall time to participate in this study is up to 18 months. Participants will make 11 visits to the clinic including a follow-up visit 6 months after the last dose of study medication.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants aged 18 to 49 years of age at the time of enrollment.
2. Are in good health at the time of entry into the trial as determined by medical history, physical examination and clinical judgment of the investigator.
3. Participants with a signed informed consent form and any required privacy authorization prior to the initiation of any trial procedures and after the nature of the trial has been explained according to local regulatory requirements.
4. Can comply with trial procedures and are available for the duration of the trial.

Exclusion Criteria:

1. Has a history of acute gastroenteritis within 14 days of enrollment.
2. Has a clinically significant active infection (as assessed by the investigator) or oral body temperature 38°C (100.4°F) or higher within 3 days of the intended date of vaccination.
3. Has received antipyretic/analgesic medications within 24 hours prior to the intended vaccine administration.
4. Has known hypersensitivity or allergy to any of the bivalent norovirus virus-like particle (VLP) vaccine components (including excipients of the investigational vaccines).
5. Has behavioral or cognitive impairment or psychiatric disease that, in the opinion of the investigator, may interfere with the participant's ability to participate in the trial.
6. Has a history of any progressive or severe neurologic disorder, seizure disorder, or neuro-inflammatory disease (e.g., Guillain-Barré syndrome).
7. Has history or any illness that, in the opinion of the investigator, might interfere with the results of the trial or pose additional risk to the participants due to participation in the trial.
8. Has known or suspected impairment/alteration of immune function including the following:

   1. Chronic use of oral steroids (Equivalent to 20 mg/day prednisone for ≥ 12 weeks / ≥2 mg/kg body weight /day for ≥ 2 weeks) within 60 days prior to Day 1 (use of inhaled, intranasal, or topical corticosteroids is allowed).
   2. Receipt of parenteral steroids (equivalent to 20 mg/day prednisone ≥ 12 weeks / ≥2 mg/kg body weight /day for ≥2 weeks) within 60 days prior to Day 1.
   3. Receipt of immunostimulants within 60 days prior to Day 1.
   4. Receipt of parenteral, epidural, or intra-articular immunoglobulin preparation, blood products, and/or plasma derivatives within 3 months prior to Day 1 or planned during the full length of the trial.
   5. Receipt of immunosuppressive therapy within 6 months prior to Day 1.
   6. Human immunodeficiency virus (HIV) infection or HIV-related disease.
   7. Heritable immunodeficiency.
9. Has abnormalities of splenic or thymic function.
10. Has a history of any autoimmune disease.
11. Has a known bleeding diathesis or any condition that may be associated with a prolonged bleeding time.
12. Has any serious chronic or progressive disease according to judgment of the investigator (e.g., neoplasm, insulin dependent diabetes, cardiac, renal, or hepatic disease).
13. Has a body mass index (BMI) greater than or equal to 35 kg/m^2 (= weight in kg / [height in meters * height in meters]).
14. Is participating in any clinical trial with another investigational product 30 days prior to first trial visit or intent to participate in another clinical trial at any time during the conduct of this trial.
15. Participants who received any inactivated vaccines within 14 days or any live vaccines for 28 days prior to enrollment in this trial.
16. Are first degree relatives of individuals involved in trial conduct.
17. Has a history of substance or alcohol abuse within the past 2 years.
18. If female, "of childbearing potential", sexually active, and has not used any of the "acceptable contraceptive methods" for at least 2 months prior to trial entry:

    1. Of childbearing potential is defined as status post onset of menarche and not meeting any of the following conditions: menopausal for at least 2 years, status after bilateral tubal ligation for at least 1 year, status after bilateral oophorectomy, or status after hysterectomy.
    2. Acceptable birth control methods are defined as 1 or more of the following:

    i. Hormonal contraceptive (such as oral, injection, transdermal patch, implant, cervical ring).

    ii. Barrier (condom with spermicide or diaphragm with spermicide) each and every time during intercourse.

    iii. Intrauterine device (IUD). iv. Monogamous relationship with vasectomized partner. Partner must have been vasectomized for at least 6 months prior to the participant's trial entry.
19. Female participants of childbearing potential and sexually active, who refuse to use an "acceptable contraceptive method" from Day 1 through 6 months after the last dose of investigational vaccine.
20. Female participants who plan to donate ova from Day 1 through 6 months after the last dose of investigational vaccine.
21. Female participants with any positive pregnancy test.
22. Female participants who are pregnant or breastfeeding.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 454 (Actual)
Dates: Start 2014-05-15 (Actual); Primary Completion 2016-01-06 (Actual); Study Completion 2016-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (10):
- United States (10):
  - California Research Foundation, San Diego, California
  - Benchmark Research San Francisco, San Francisco, California
  - Clin Research of South Florida, Coral Gables, Florida
  - SNBL, Baltimore, Maryland
  - St. Louis University, School of Medicine, St Louis, Missouri
  - Rochester Clinical Research, Rochester, New York
  - University of Rochester, Rochester, New York
  - Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio
  - Benchmark Research Austin, Austin, Texas
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- [Derived] Atmar RL, Baehner F, Cramer JP, Lloyd E, Sherwood J, Borkowski A, Mendelman PM; NOR-201 Study Group. Persistence of Antibodies to 2 Virus-Like Particle Norovirus Vaccine Candidate Formulations in Healthy Adults: 1-Year Follow-up With Memory Probe Vaccination. J Infect Dis. 2019 Jul 19;220(4):603-614. doi: 10.1093/infdis/jiz170. PMID 31001633
- [Derived] Atmar RL, Baehner F, Cramer JP, Song E, Borkowski A, Mendelman PM; NOR-201 Study Group. Rapid Responses to 2 Virus-Like Particle Norovirus Vaccine Candidate Formulations in Healthy Adults: A Randomized Controlled Trial. J Infect Dis. 2016 Sep 15;214(6):845-53. doi: 10.1093/infdis/jiw259. Epub 2016 Jun 28. PMID 27354368

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 10 investigative sites in the United States from 28 April 2014 to 14 January 2016.
Pre-assignment Details: Healthy volunteers were enrolled equally in 1 of 3 norovirus bivalent virus like particle (VLP) vaccine unique formulation treatment groups to receive: 2 formulation arms received 2 doses and 1 formulation arm received 1 dose.
Groups:
- Saline Placebo + GI.1/GII.4 15/15 μg (No MPL): Intramuscular (IM) saline placebo on Day 1, followed by IM norovirus bivalent virus like particle (VLP) vaccine (15 µg of GI.1 norovirus VLP and 15 µg GII.4 norovirus VLP) adjuvanted with 500 µg aluminum hydroxide (no monophosphoryl lipid A [MPL]), on Day 365.
- GI.1/GII.4 15/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL): IM norovirus bivalent VLP vaccine (15 µg of GI.1 norovirus VLP and 50 µg GII.4 norovirus VLP) adjuvanted with 50 µg MPL and 500 µg aluminum hydroxide, on Day 1, followed by IM norovirus bivalent VLP vaccine (15 µg of GI.1 norovirus VLP and 15 µg GII.4 norovirus VLP) adjuvanted with 500 µg aluminum hydroxide, (no MPL) on Day 365.
- GI.1/GII.4 50/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL): IM norovirus bivalent VLP vaccine (50 µg of GI.1 norovirus VLP and 50 µg GII.4 norovirus VLP) adjuvanted with 50 µg MPL and 500 µg aluminum hydroxide, on Day 1, followed by IM norovirus bivalent VLP vaccine (15 µg of GI.1 norovirus VLP and 15 µg GII.4 norovirus VLP) adjuvanted with 500 µg aluminum hydroxide (no MPL), on Day 365.
Period: Overall Study
Arm/Group | Saline Placebo + GI.1/GII.4 15/15 μg (No MPL) | GI.1/GII.4 15/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL) | GI.1/GII.4 50/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL)
Started | 153 | 147 | 154
Randomized and Received Treatment | 153 | 145 | 154
Received Booster (Second Vaccination) | 126 | 109 | 116
Completed | 122 | 105 | 111
Not Completed | 31 | 42 | 43
Not completed — Protocol Violation | 2 | 1 | 2
Not completed — Adverse Event | 2 | 3 | 4
Not completed — Lost to Follow-up | 12 | 19 | 17
Not completed — Withdrawal by Subject | 7 | 9 | 11
Not completed — Pregnancy | 4 | 4 | 2
Not completed — Physician Decision | 0 | 1 | 3
Not completed — Reason Not Specified | 4 | 5 | 4

BASELINE CHARACTERISTICS:
Population: Randomized Set included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Saline Placebo + GI.1/GII.4 15/15 μg (No MPL) | GI.1/GII.4 15/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL) | GI.1/GII.4 50/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL) | Total
Number analyzed (Participants) | 153 | 147 | 154 | 454
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.9 (8.87) | 33.4 (9.26) | 34.0 (8.78) | 33.5 (8.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 89 | 75 | 253
  Male | 64 | 58 | 79 | 201
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 34 | 38 | 46 | 118
  Non-Hispanic and Latino | 117 | 109 | 107 | 333
  Not Reported | 1 | 0 | 1 | 2
  Unknown | 1 | 0 | 0 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 | 2 | 2
  Asian | 5 | 3 | 2 | 10
  Black or African American | 41 | 49 | 47 | 137
  Native Hawaiian or Other Pacific Islander | 3 | 2 | 2 | 7
  White | 100 | 91 | 94 | 285
  Other | 1 | 1 | 2 | 4
  Multiracial | 3 | 1 | 5 | 9
Region of Enrollment [Number; unit: participants]
  United States | 153 | 147 | 154 | 454
Height [Mean (Standard Deviation); unit: cm] | 169.91 (9.228) | 168.89 (9.670) | 171.24 (9.859) | 170.03 (9.616)
Weight [Mean (Standard Deviation); unit: kg] | 76.50 (14.924) | 75.56 (14.720) | 76.91 (15.598) | 76.33 (15.068)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.40 (4.125) | 26.44 (4.427) | 26.14 (4.313) | 26.32 (4.281)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Solicited Local Adverse Events (AEs) at Injection Site After the First Injection
Description: Solicited local AEs at injection site are defined as: pain, erythema, induration, and swelling that occurred within 7 days after the primary injection.
Time Frame: Days 1 through 7
Population: Safety Analysis Set included all participants who received at least one dose of trial vaccination.
Measure: Number; unit: percentage of participants
Arm/Group | Saline Placebo + GI.1/GII.4 15/15 μg (No MPL) | GI.1/GII.4 15/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL) | GI.1/GII.4 50/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL)
Number analyzed (Participants) | 153 | 145 | 154
percentage of participants
  Any Solicited Local AEs | 7.8 | 64.1 | 72.7
  Pain | 7.8 | 64.1 | 72.7
  Erythema | 0 | 0 | 0.6
  Induration | 0 | 1.4 | 1.3
  Swelling | 0 | 2.1 | 0.6

2. Primary Outcome: Percentage of Participants With Solicited Systemic Adverse Events (AEs) After the First Injection
Description: Solicited systemic AEs are defined as: headache, fatigue, myalgia, arthralgia, vomiting, and diarrhea that occurred within 7 days after the primary injection.
Time Frame: Days 1 through 7
Population: Safety Analysis Set included all participants who received at least one dose of trial vaccination.
Measure: Number; unit: percentage of participants
Arm/Group | Saline Placebo + GI.1/GII.4 15/15 μg (No MPL) | GI.1/GII.4 15/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL) | GI.1/GII.4 50/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL)
Number analyzed (Participants) | 153 | 145 | 154
percentage of participants
  Any Solicited Systemic AEs | 26.8 | 33.1 | 45.5
  Headache | 16.3 | 15.9 | 18.2
  Fatigue | 17.0 | 15.9 | 16.2
  Myalgia | 7.2 | 19.3 | 25.3
  Arthralgia | 3.3 | 4.8 | 7.8
  Vomiting | 1.3 | 1.4 | 1.9
  Diarrhea | 7.8 | 7.6 | 10.4

3. Primary Outcome: Percentage of Participants With Elevated Daily Oral Temperature (Fever) After the First Injection
Description: Fever is defined as greater than or equal to 38°C (100.4°F). Oral body temperature measurement was performed using the thermometer provided by the site for 7 days after each injection. The highest body temperature observed each day was recorded on the Diary Card also provided by the site.
Time Frame: Days 1 through 7
Population: Safety Analysis Set included all participants who received at least one dose of trial vaccination.
Measure: Number; unit: percentage of participants
Arm/Group | Saline Placebo + GI.1/GII.4 15/15 μg (No MPL) | GI.1/GII.4 15/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL) | GI.1/GII.4 50/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL)
Number analyzed (Participants) | 153 | 145 | 154
percentage of participants | 0 | 0.7 | 0

4. Primary Outcome: Percentage of Participants With Unsolicited Adverse Events (AEs) After the First Injection
Description: Unsolicited AEs are any AEs that are not solicited local or systemic AEs, as defined by this study.
Time Frame: Days 1 through 28
Population: Safety Analysis Set included all participants who received at least one dose of trial vaccination.
Measure: Number; unit: percentage of participants
Arm/Group | Saline Placebo + GI.1/GII.4 15/15 μg (No MPL) | GI.1/GII.4 15/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL) | GI.1/GII.4 50/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL)
Number analyzed (Participants) | 153 | 145 | 154
percentage of participants | 23.5 | 16.6 | 21.4

5. Primary Outcome: Percentage of Participants With Serious Adverse Events (SAEs) After the First Injection
Description: A serious adverse event (SAE) is any untoward medical occurrence or effect that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability / incapacity, is a congenital anomaly / birth defect or is medically important due to other reasons than the above mentioned criteria.
Time Frame: From first injection (Day 1) to second injection pre-dose (Up to Day 365)
Population: Safety Analysis Set included all participants who received at least one dose of trial vaccination.
Measure: Number; unit: percentage of participants
Arm/Group | Saline Placebo + GI.1/GII.4 15/15 μg (No MPL) | GI.1/GII.4 15/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL) | GI.1/GII.4 50/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL)
Number analyzed (Participants) | 153 | 145 | 154
percentage of participants | 1.3 | 2.1 | 3.2

6. Primary Outcome: Percentage of Participants With Serious Adverse Events (SAEs) After the Second Injection
Description: as for outcome 5
Time Frame: From second injection (Day 365) to 6 months after second injection (Up to Day 545)
Population: Participants from the Safety Analysis Set who received a second injection.
Measure: Number; unit: percentage of participants
Arm/Group | Saline Placebo + GI.1/GII.4 15/15 μg (No MPL) | GI.1/GII.4 15/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL) | GI.1/GII.4 50/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL)
Number analyzed (Participants) | 126 | 109 | 116
percentage of participants | 1.6 | 0.9 | 0.9

7. Primary Outcome: Percentage of Participants With Adverse Events of Special Interest (AESI) After the First Injection
Description: AESIs are AEs that are not solicited local or systemic AEs, they are predefined AEs that required close monitoring and prompt reporting to the sponsor. AESI included protocol specified Cardiac Disorders, Gastrointestinal Disorders, Immune System Disorders, Infections and Infestations, Musculoskeletal and Connective Tissue Diseases, Neuroinflammatory Disorders, Renal and Urinary Disorders, Skin Disorders, Thyroid Disorders, Vascular Disorders and Other Disorders.
Time Frame: From first injection (Day 1) to second injection pre-dose (Up to Day 365)
Population: Safety Analysis Set included all participants who received at least one dose of trial vaccination.
Measure: Number; unit: percentage of participants
Arm/Group | Saline Placebo + GI.1/GII.4 15/15 μg (No MPL) | GI.1/GII.4 15/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL) | GI.1/GII.4 50/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL)
Number analyzed (Participants) | 153 | 145 | 154
percentage of participants | 1.3 | 2.1 | 1.3

8. Primary Outcome: Percentage of Participants With Adverse Events of Special Interest (AESI) After the Second Injection
Description: as for outcome 7
Time Frame: From second injection (Day 365) to 6 months after second injection (Up to Day 545)
Population: Participants from the Safety Analysis Set who received a second injection.
Measure: Number; unit: percentage of participants
Arm/Group | Saline Placebo + GI.1/GII.4 15/15 μg (No MPL) | GI.1/GII.4 15/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL) | GI.1/GII.4 50/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL)
Number analyzed (Participants) | 126 | 109 | 116
percentage of participants | 3.2 | 0 | 0.9

9. Primary Outcome: Percentage of Participants With Any Adverse Event (AE) Leading to Withdrawal From the Study
Description: Withdrawal due to an AE occurred if the participant experienced an AE that required early termination because continued participation imposed an unacceptable risk to the participant's health or the participant was unwilling to continue because of the AE.
Time Frame: Unsolicited AEs 28 days after each injection (Days 1 to 28 and Days 365 to 393), and Serious Adverse Events (SAEs) throughout the trial (Up to Day 545)
Population: Safety Analysis Set included all participants who received at least one dose of trial vaccination.
Measure: Number; unit: percentage of participants
Arm/Group | Saline Placebo + GI.1/GII.4 15/15 μg (No MPL) | GI.1/GII.4 15/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL) | GI.1/GII.4 50/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL)
Number analyzed (Participants) | 153 | 145 | 154
percentage of participants | 1.3 | 1.4 | 2.6

10. Secondary Outcome: Percentage of Participants With Solicited Local Adverse Events (AEs) at Injection Site After the Second Injection
Description: Solicited local AEs at injection site are defined as: pain, erythema, induration, and swelling that occurred within 7 days after the vaccination on Day 365.
Time Frame: Days 365 through 371
Population: Participants from the Safety Analysis Set who received a second injection.
Measure: Number; unit: percentage of participants
Arm/Group | Saline Placebo + GI.1/GII.4 15/15 μg (No MPL) | GI.1/GII.4 15/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL) | GI.1/GII.4 50/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL)
Number analyzed (Participants) | 126 | 109 | 116
percentage of participants
  Any Solicited Local AEs | 41.3 | 41.3 | 44.0
  Pain | 41.3 | 41.3 | 44.0
  Erythema | 0.8 | 0.9 | 0
  Induration | 0 | 0 | 0
  Swelling | 0 | 2.8 | 0

11. Secondary Outcome: Percentage of Participants With Solicited Systemic Adverse Events (AEs) After the Second Injection
Description: Solicited systemic AEs are defined as: headache, fatigue, myalgia, arthralgia, vomiting, and diarrhea that occurred within 7 days after the vaccination on Day 365.
Time Frame: Days 365 through 371
Population: Participants from the Safety Analysis Set who received a second injection.
Measure: Number; unit: percentage of participants
Arm/Group | Saline Placebo + GI.1/GII.4 15/15 μg (No MPL) | GI.1/GII.4 15/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL) | GI.1/GII.4 50/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL)
Number analyzed (Participants) | 126 | 109 | 116
percentage of participants
  Any Solicited Systemic AEs | 28.6 | 25.7 | 31.9
  Headache | 11.9 | 11.0 | 14.7
  Fatigue | 11.1 | 14.7 | 17.2
  Myalgia | 15.1 | 15.6 | 14.7
  Arthralgia | 0.8 | 7.3 | 6.0
  Vomiting | 2.4 | 1.8 | 1.7
  Diarrhea | 4.0 | 7.3 | 8.6

12. Secondary Outcome: Percentage of Participants With Elevated Daily Oral Temperature (Fever) After the Second Injection
Description: Fever is defined as greater than or equal to 38°C (100.4°F). Oral body temperature measurement was performed using the thermometer provided by the site for 7 days after each vaccination. The highest body temperature observed each day was recorded on the Diary Card also provided by the site.
Time Frame: Days 365 through 371
Population: Participants from the Safety Analysis Set who received a second injection.
Measure: Number; unit: percentage of participants
Arm/Group | Saline Placebo + GI.1/GII.4 15/15 μg (No MPL) | GI.1/GII.4 15/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL) | GI.1/GII.4 50/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL)
Number analyzed (Participants) | 126 | 109 | 116
percentage of participants | 0 | 0.9 | 2.6

13. Secondary Outcome: Percentage of Participants With Unsolicited Adverse Events (AEs) After the Second Injection
Description: Unsolicited AEs are any AEs that are not solicited local or systemic AEs, as defined by this study.
Time Frame: Days 365 through 393
Population: Participants from the Safety Analysis Set who received a second injection.
Measure: Number; unit: percentage of participants
Arm/Group | Saline Placebo + GI.1/GII.4 15/15 μg (No MPL) | GI.1/GII.4 15/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL) | GI.1/GII.4 50/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL)
Number analyzed (Participants) | 126 | 109 | 116
percentage of participants | 20.6 | 14.7 | 14.7

14. Secondary Outcome: Percentage of Participants With a Seroresponse in Both Serum Anti-norovirus GI.1 VLP and GII.4 VLP (Pan-Ig ELISA)
Description: Seroresponse is defined as 4-fold rise or greater in serum anti-norovirus antibody titers for both GI.1 virus-Like particle (VLP) and GII.4 VLP as measured by pan immunoglobulin (Pan-Ig) enzyme-linked immunosorbent assay (ELISA).
Time Frame: Baseline and Day 28
Population: Per Protocol Set included all participants in Full Analysis Set, who had evaluable blood samples at baseline, and Day 28 within the specified window (+/- 7 days), and did not have major protocol violations.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Saline Placebo + GI.1/GII.4 15/15 μg (No MPL) | GI.1/GII.4 15/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL) | GI.1/GII.4 50/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL)
Number analyzed (Participants) | 151 | 140 | 151
percentage of participants | 2.6 [0.7 to 6.6] | 70.7 [62.4 to 78.1] | 64.9 [56.7 to 72.5]

15. Secondary Outcome: Percentage of Participants With a Seroresponse in Serum Anti-norovirus GI.1 VLP (Pan-Ig ELISA)
Description: Seroresponse is defined as 4-fold rise or greater in serum anti-norovirus antibody titers for GI.1 virus-Like particle (VLP) as measured by pan immunoglobulin (Pan-Ig) enzyme-linked immunosorbent assay (ELISA).
Time Frame: Baseline and Day 28
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Saline Placebo + GI.1/GII.4 15/15 μg (No MPL) | GI.1/GII.4 15/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL) | GI.1/GII.4 50/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL)
Number analyzed (Participants) | 151 | 140 | 151
percentage of participants | 8.6 [4.7 to 14.3] | 91.4 [85.5 to 95.5] | 90.1 [84.1 to 94.3]

16. Secondary Outcome: Percentage of Participants With a Seroresponse in Serum Anti-norovirus GII.4 VLP (Pan-Ig ELISA)
Description: Seroresponse is defined as 4-fold rise or greater in serum anti-norovirus antibody titers for GII.4 virus-like particles (VLP) as measured by pan immunoglobulin (Pan-Ig) enzyme-linked immunosorbent assay (ELISA).
Time Frame: Baseline and Day 28
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Saline Placebo + GI.1/GII.4 15/15 μg (No MPL) | GI.1/GII.4 15/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL) | GI.1/GII.4 50/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL)
Number analyzed (Participants) | 151 | 140 | 151
percentage of participants | 4.6 [1.9 to 9.3] | 75.0 [67.0 to 81.9] | 69.5 [61.5 to 76.8]

17. Secondary Outcome: Geometric Mean Titer (GMT) of GI.1 VLP Antibody Titers (Pan-Ig ELISA)
Description: Geometric mean titer (GMT) of anti-norovirus GI.1 VLP antibody titers as measured by Pan-Ig ELISA.
Time Frame: Day 28
Population: as for outcome 14
Measure: Geometric Mean (Standard Deviation); unit: titer
Arm/Group | Saline Placebo + GI.1/GII.4 15/15 μg (No MPL) | GI.1/GII.4 15/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL) | GI.1/GII.4 50/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL)
Number analyzed (Participants) | 151 | 140 | 151
titer | 366.8 (6.29) | 13023.2 (3.40) | 18711.8 (3.84)

18. Secondary Outcome: Geometric Mean Titer (GMT) of GII.4 VLP Antibody Titers (Pan-Ig ELISA)
Description: Geometric mean titer (GMT) of anti-norovirus GII.4 VLP antibody titers as measured by Pan-Ig ELISA.
Time Frame: Day 28
Population: as for outcome 14
Measure: Geometric Mean (Standard Deviation); unit: titer
Arm/Group | Saline Placebo + GI.1/GII.4 15/15 μg (No MPL) | GI.1/GII.4 15/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL) | GI.1/GII.4 50/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL)
Number analyzed (Participants) | 151 | 140 | 151
titer | 955.5 (5.08) | 11275.5 (2.38) | 8667.9 (2.84)

19. Secondary Outcome: Geometric Mean Fold Rise (GMFR) of GI.1 VLP Antibody Titers (Pan-Ig ELISA)
Description: Geometric mean fold rise (GMFR) of anti-norovirus GI.1 VLP antibody titers as measured by Pan-Ig ELISA.
Time Frame: Day 28
Population: as for outcome 14
Measure: Geometric Mean (Standard Deviation); unit: ratio
Arm/Group | Saline Placebo + GI.1/GII.4 15/15 μg (No MPL) | GI.1/GII.4 15/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL) | GI.1/GII.4 50/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL)
Number analyzed (Participants) | 151 | 140 | 151
ratio | 1.3 (3.81) | 37.6 (6.11) | 55.9 (5.90)

20. Secondary Outcome: Geometric Mean Fold Rise (GMFR) of GII.4 VLP Antibody Titers (Pan-Ig ELISA)
Description: Geometric mean fold rise (GMFR) of anti-norovirus GII.4 VLP antibody titers as measured by Pan-Ig ELISA.
Time Frame: Day 28
Population: as for outcome 14
Measure: Geometric Mean (Standard Deviation); unit: ratio
Arm/Group | Saline Placebo + GI.1/GII.4 15/15 μg (No MPL) | GI.1/GII.4 15/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL) | GI.1/GII.4 50/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL)
Number analyzed (Participants) | 151 | 140 | 151
ratio | 1.1 (2.08) | 10.7 (4.35) | 7.4 (3.46)

21. Secondary Outcome: Percentage of Participants With a Seroresponse in Both Serum Anti-norovirus GI.1 VLP and GII.4 VLP (HBGA)
Description: Seroresponse is defined as 4-fold rise or greater in serum anti-norovirus antibody titers for both GI.1 virus-Like particle (VLP) and GII.4 VLP as measured by histoblood group antigen (HBGA) binding assay.
Time Frame: Baseline and Day 28
Population: Participants from the Per Protocol Set, all participants in Full Analysis Set, who had evaluable blood samples at baseline, and Day 28 within the specified window (+/- 7 days), and did not have major protocol violations, with data available for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Saline Placebo + GI.1/GII.4 15/15 μg (No MPL) | GI.1/GII.4 15/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL) | GI.1/GII.4 50/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL)
Number analyzed (Participants) | 151 | 139 | 151
percentage of participants | 2.0 [0.4 to 5.7] | 55.4 [46.7 to 63.8] | 55.0 [46.7 to 63.1]

22. Secondary Outcome: Percentage of Participants With a Seroresponse in Serum GI.1 VLP Antibody Titers (HBGA)
Description: Seroresponse is defined as 4-fold rise or greater in serum anti-norovirus antibody titers for GI.1 virus-Like particle (VLP) as measured by HBGA binding assay.
Time Frame: Baseline and Day 28
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Saline Placebo + GI.1/GII.4 15/15 μg (No MPL) | GI.1/GII.4 15/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL) | GI.1/GII.4 50/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL)
Number analyzed (Participants) | 151 | 140 | 151
percentage of participants | 3.3 [1.1 to 7.6] | 74.3 [66.2 to 81.3] | 80.8 [73.6 to 86.7]

23. Secondary Outcome: Percentage of Participants With a Seroresponse in Serum GII.4 VLP Antibody Titers (HBGA)
Description: Seroresponse is defined as 4-fold rise or greater in serum anti-norovirus antibody titers for GII.4 virus-Like particle (VLP) as measured by HBGA binding assay.
Time Frame: Baseline and Day 28
Population: Participants from the Per Protocol Set, all participants in Full Analysis Set, who had evaluable blood samples at baseline, and Day 28 within the specified window (+/- 7 days), and did not have major protocol violations, with data for this outcome measure
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Saline Placebo + GI.1/GII.4 15/15 μg (No MPL) | GI.1/GII.4 15/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL) | GI.1/GII.4 50/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL)
Number analyzed (Participants) | 151 | 139 | 151
percentage of participants | 2.6 [0.7 to 6.6] | 71.2 [62.9 to 78.6] | 68.2 [60.1 to 75.5]

24. Secondary Outcome: Blocking Titers 50 (BT50) of Anti-Norovirus GI.1 VLP Antibody Titers (HBGA)
Description: Blocking titers 50 (BT50) of anti-norovirus GI.1 VLP antibody titers as measured by HBGA binding assay.
Time Frame: Day 28
Population: as for outcome 14
Measure: Geometric Mean (Standard Deviation); unit: titer
Arm/Group | Saline Placebo + GI.1/GII.4 15/15 μg (No MPL) | GI.1/GII.4 15/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL) | GI.1/GII.4 50/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL)
Number analyzed (Participants) | 151 | 140 | 151
titer | 20.7 (2.38) | 170.9 (3.90) | 207.8 (3.94)

25. Secondary Outcome: Blocking Titers 50 (BT50) of Anti-Norovirus GII.4 VLP Antibody Titers (HBGA)
Description: Blocking titers 50 (BT50) of anti-norovirus GII.4 VLP antibody titers as measured by HBGA binding assay.
Time Frame: Day 28
Population: as for outcome 21
Measure: Geometric Mean (Standard Deviation); unit: titer
Arm/Group | Saline Placebo + GI.1/GII.4 15/15 μg (No MPL) | GI.1/GII.4 15/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL) | GI.1/GII.4 50/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL)
Number analyzed (Participants) | 151 | 139 | 151
titer | 80.1 (4.33) | 804.3 (3.32) | 631.3 (3.05)

26. Secondary Outcome: Geometric Mean Fold Rise (GMFR) of GI.1 VLP Antibody Titers (HBGA)
Description: Geometric mean fold rise (GMFR) of anti-norovirus GI.1 VLP antibody titers as measured by HBGA binding assay.
Time Frame: Day 28
Population: as for outcome 14
Measure: Geometric Mean (Standard Deviation); unit: ratio
Arm/Group | Saline Placebo + GI.1/GII.4 15/15 μg (No MPL) | GI.1/GII.4 15/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL) | GI.1/GII.4 50/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL)
Number analyzed (Participants) | 151 | 140 | 151
ratio | 1.1 (1.69) | 8.9 (3.64) | 10.5 (3.56)

27. Secondary Outcome: Geometric Mean Fold Rise (GMFR) of GII.4 VLP Antibody Titers (HBGA)
Description: Geometric mean fold rise (GMFR) of anti-norovirus GII.4 VLP antibody titers as measured by the HBGA binding assay.
Time Frame: Day 28
Population: as for outcome 21
Measure: Geometric Mean (Standard Deviation); unit: ratio
Arm/Group | Saline Placebo + GI.1/GII.4 15/15 μg (No MPL) | GI.1/GII.4 15/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL) | GI.1/GII.4 50/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL)
Number analyzed (Participants) | 151 | 139 | 151
ratio | 1.0 (1.77) | 9.7 (4.03) | 7.3 (3.23)

ADVERSE EVENTS:
Time Frame: Unsolicited AEs 28 days after each injection (Days 1 to 28 and Days 365 to 393), and Serious Adverse Events (SAEs) throughout the trial (Up to Day 545)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Saline Placebo + GI.1/GII.4 15/15 μg (No MPL) | GI.1/GII.4 15/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL) | GI.1/GII.4 50/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL)
Serious Adverse Events (participants affected / at risk) | 4/153 | 4/145 | 6/154
Other Adverse Events (participants affected / at risk) | 33/153 | 24/145 | 25/154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Saline Placebo + GI.1/GII.4 15/15 μg (No MPL) (N=153) | GI.1/GII.4 15/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL) (N=145) | GI.1/GII.4 50/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL) (N=154)
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0
Basedow's disease (Endocrine disorders) | 0 | 0 | 1
Retinal detachment (Eye disorders) | 1 | 0 | 0
Injection site pain (General disorders) | 0 | 0 | 1
Kidney infection (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 1 | 0
Neuralgic amyotrophy (Nervous system disorders) | 0 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 1 | 1
Depression (Psychiatric disorders) | 0 | 1 | 1
Post-traumatic stress disorder (Psychiatric disorders) | 0 | 0 | 1
Schizophrenia (Psychiatric disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Saline Placebo + GI.1/GII.4 15/15 μg (No MPL) (N=153) | GI.1/GII.4 15/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL) (N=145) | GI.1/GII.4 50/50 μg - MPL 50 μg + GI.1/GII.4 15/15 μg (no MPL) (N=154)
Nausea (Gastrointestinal disorders) | 7 | 3 | 5
Diarrhoea (Gastrointestinal disorders) | 3 | 4 | 3
Abdominal pain upper (Gastrointestinal disorders) | 3 | 3 | 1
Fatigue (General disorders) | 2 | 1 | 4
Injection site bruising (General disorders) | 4 | 1 | 0
Injection site pain (General disorders) | 0 | 3 | 1
Nasopharyngitis (Infections and infestations) | 2 | 4 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 5 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0 | 4
Headache (Nervous system disorders) | 11 | 5 | 10
Dizziness (Nervous system disorders) | 2 | 3 | 1
Sinus headache (Nervous system disorders) | 2 | 0 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.